CLINICAL TRIAL: NCT02786056
Title: Feasibility of Regional Lung Ventilation Imaging Using 3T MR Imaging With Ultrashort Echo Time (UTE) Pulse Sequences (PULMOREM Study)
Brief Title: Feasibility of Regional Lung Ventilation Imaging Using 3T MR Imaging With Ultrashort Echo Time (UTE) Pulse Sequences
Acronym: PULMOREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2014_843_0011
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Magnetic Resonance Imaging
Keywords: Respiratory Function Tests; Lung

ARMS (1):
- Lung MRI examination (Experimental)
  Interventions: Other: Lung MRI examination

INTERVENTIONS:
Other: Lung MRI examination — Lung MRI examination is performed for approximately 30 min on a 3T machine (Achieva 3T, Philips) using UTE sequences, both during free breathing with image synchronisation using an echo-navigator, and during an end-inspiratory and end-expiratory pauses. In the 10 first subjects, the MR protocol is optimized in order to maximize MRI parenchymal signal intensity, signal-to-noise ratio and contrast-to-noise ratio. The final image acquisition parameters will be applied in the following 30 subjects in order to assess the outcomes of the study.

SUMMARY:
Structural lung and airway alterations in CF lead to focal or heterogeneous abnormalities in regional lung ventilation. The quantitative assessment of structural and functional alterations in the lung is of great importance for the phenotyping and follow-up of CF patients. The goal of this study is to assess the feasibility of measuring the changes in proton density in the lung parenchyma with inflation and deflation during the respiratory cycle, using ultrashort echo time (UTE) pulse sequence MRI, in healthy adult volunteers.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common severe autosomal recessive genetic disease in Caucasians. severe structural alterations in the airways and parenchyma, such as bronchiectasis, mucus plugging, air trapping and infiltrations. These in turn result in focal or heterogeneous abnormalities in regional lung ventilation. End-stage lung disease remains the main cause of morbidity and mortality in CF patients. Currently, new targeted CFTR correctors and potentiators are under trial. The quantitative assessment of structural and functional alterations in the lung is of great importance for the phenotyping and follow-up of CF patients, and for the assessment of targeted therapeutic interventions. Computed tomography (CT) is considered as the technology of choice for lung imaging in CF. However, CT requires exposure to significant ionizing radiation, which is a major concern in the pediatric population because children are more radiosensitive than adults and there is an increased risk of radiation-induced cancer from the cumulative dose related to repeated CT investigations. Recent improvements in magnetic resonance imaging (MRI) technology offer a non-ionizing alternative to CT for imaging the lung parenchyma. The goal of this study is to assess the feasibility of measuring the changes in proton density in the lung parenchyma with inflation and deflation during the respiratory cycle, using ultrashort echo time (UTE) pulse sequence MRI, in healthy adult volunteers. If the regional changes in proton density in the lung parenchyma during the respiratory cycle prove to be measurable in healthy volunteers, then MRI can be used to quantify regional lung ventilation. This would offer a unique non-invasive, radiation- and contrast media-free alternative to CT for phenotyping and follow-up of CF patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 to 65 years.
* Written informed consent.
* Health insurance policy holder.

Exclusion Criteria:

* Current smoker
* Detained or legally irresponsable.
* No social security or health insurance policy.
* Chronic respiratory diseases (such as asthma, COPD, CF, pulmonary fibrosis or hypertension).
* Acute or recent lower respiratory tract infection.
* Smoking or heavy meal less than 1 hour prior to imaging.
* Acute or recent serious health condition (such as : myocardial infarction, pulmonary embolism…).
* MRI contraindications: Magnetically activated implanted devices (cardiac pacemakers, insulin pumps, neurostimulators, cochlear implants), metal inside the eye or the brain (aneurysm clip, metallic ocular foreign body), cardiac valvular prosthesis (Starr-Edwards pre-6000), subject with claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Correlation between the magnitude of change in MRI signal intensity from end-inspiration to end-expiration, averaged over the entire 3D lung image, and tidal volume measured by spirometry during imaging | 30 days

SECONDARY OUTCOMES:
Agreement between the correlation coefficient of MRI signal intensity change vs. tidal volume acquired during free breathing, and that acquired in static conditions (end-inspiration, end-expiration) | 30 days
Comparison of signal-to-noise and contrast-to-noise ratio of lung parenchyma measured using UTE MRI to values published in the litterature. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu GUILBART, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France